CLINICAL TRIAL: NCT01046864
Title: A Phase Ib Multiple Ascending Dose Study to Evaluate the Safety of Brivanib in Combination With 5-Fluorouracil/Leucovorin (5FU/LV) and Brivanib in Combination With 5-Fluorouracil/Leucovorin/Irinotecan (FOLFIRI) in Subjects With Advanced or Metastatic Gastrointestinal Malignancies
Brief Title: Combination of Brivanib With 5-Fluorouracil/Leucovorin (5FU/LV) and 5-Fluorouracil/Leucovorin/Irinotecan (FOLFIRI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CA182-046; 2009-016699-63 (EudraCT Number)
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Gastro-Intestinal Cancer
Keywords: Gastro-Intestinal Cancer, NOS
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — Fluorouracil; Leucovorin; Irinotecan; brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: 5-FU; Drug: Leucovorin; Drug: Brivanib
- Arm 2 (Experimental)
  Interventions: Drug: 5-FU; Drug: Leucovorin; Drug: Irinotecan; Drug: Brivanib
- Arm 3 (Experimental): Japanese Population
  Interventions: Drug: 5-FU; Drug: Leucovorin; Drug: Irinotecan; Drug: Brivanib

INTERVENTIONS:
Drug: 5-FU — IV solution, IV bolus over 2-4 minutes, 400 mg/m², Every 14 days, Until disease progression/toxicity
  Other Names: Fluorouracil
Drug: Leucovorin — IV solution, IV over 2 hours, 400 mg/m², Every 14 days, Until disease progression/toxicity
  Other Names: Folinic acid
Drug: 5-FU — IV solution, IV infusion over 46 hours, 2400 mg/m², Every 14 days, Until disease progression/toxicity
  Other Names: Fluorouracil
Drug: Irinotecan — IV solution, IV over 90 minutes, 180 mg/m², Every 14 days, Until disease progression/toxicity
  Other Names: Camptosar
  Arms: Arm 2; Arm 3
Drug: Brivanib — Tablets, Oral, 400 - 800 mg, once daily, Until disease progression/toxicity
  Arms: Arm 1
Drug: Brivanib — Tablets, Oral, 600 - 800 mg, once daily, Until disease progression/toxicity
  Other Names: BMS-582664
  Arms: Arm 2
Drug: Brivanib — Tablets, Oral, 800 mg, once daily, Until disease progression/toxicity
  Other Names: BMS-582664
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine a safe and maximum tolerable dose of Brivanib when combined with standard dose 5FU/LV and FOLFIRI.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological/cytological confirmed diagnosis of Gastrointestinal malignancy, except pancreatic cancer
* Eligible for 5FU/LV or FOLFIRI chemotherapy
* ECOG 0-1
* Able to swallow and tolerate tablets
* Life expectancy of 3 months

Exclusion Criteria:

* Unwilling to use acceptable method to avoid pregnancy of partner/self for the entire study period and up to 4 weeks after last dose
* Women who are pregnant or breastfeeding
* Pancreatic cancer
* Known brain metastasis, evidence of leptomeningeal disease
* History of thrombo-embolic disease
* Hemorrhage/bleeding events
* Uncontrolled or significant cardiovascular disease
* Any 3 or more of the following risk factors: arterial thrombosis , smoking, hypercholesterolemia, hypertension, obesity (BMS>30) and diabetes
* Pre-existing thyroid abnormality, not maintained with medication
* QTC (Fridericia) >450 msec on two consecutive ECG's
* Subjects with concomitant second malignancies ( except adequately treated non-melanoma skin, in situ carcinoma of bladder, cervix or breast, early prostate cancer)
* Any major surgery within 4 weeks of study drug administration
* Increased levels of both D-Dimer and Prothrombin fragment 1 +2
* Arm B and C only-positive UGT1A1 genotype of TA7/TA7
* History of allergy of brivanib or drug class
* History of severe reactions to fluoropyrimidine therapy or irinotecan
* Prior therapy with brivanib

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety-Toxicity, evaluated according to NCI Common Terminology Criteria for Adverse Events v3.0. Assessments based on medical review of adverse events, results of vital signs, ECGs, echocardiography, physical examinations, and clinical laboratory tests | Cycle 4, Day 1

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax, Tmax, AUC (TAU), T-HALF) plasma concentration vs time for brivanib given alone and in combination with FOLFIRI. Individual concentrations (C) of 5FU will be calculated from samples on Day 2 in the presence and absence of Brivanib | Cycle 2, Day 2
Efficacy-Tumor BOR determined for treated subjects by radiological responses assessed by CT scan or MRI, by RECIST criteria (v1.1). Radiological tumor assessments to evaluate response & progression will be done every 8 wks or more frequently if indicated | Every 8 weeks
Exploratory Measures (Biomarkers for Predictive Analysis): Potential predictive markers, including activity of FGF, VEGF and related pathways as well as K-RAS mutation status, will be evaluated based on blood or tumor samples | Cycle 1, Cycle 2, every other cycle

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (3):
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - Texas Oncology, Dallas, Texas
  - Scott & White Memorial Hospital And Clinic, Temple, Texas
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ottawa, Ontario
- Local Institution, Villejuif, France

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx